CLINICAL TRIAL: NCT02699255
Title: A Single-center Observational Study to Examine the Occurrence of Ventricular Arrhythmias After Pulmonary Vein Isolation
Brief Title: Ventricular Arrhythmias After Pulmonary Vein Isolation
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian Meyer, Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: WF-01/16
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2018-10

CONDITIONS: Ventricular Arrhythmias; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators study aimed to observe the occurrence of new premature ventricular complexes and other ventricular arrhythmias after pulmonary vein isolation.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common arrhythmia with a lifetime risk for development of over 20%. Pulmonary vein isolation is now established as therapy of choice for patients with symptomatic atrial fibrillation. It is well known that this interventional therapy inevitably modulates the intracardiac autonomic nervous system. While this ablation might alter atrial electrophysiology beneficially, the impact on ventricular electrophysiology remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Paroxysmal atrial fibrillation scheduled to undergo pulmonary vein isolation

Exclusion Criteria:

* Age < 18 years
* Persistent atrial fibrillation
* Life expectancy less than 12 months
* Acute myocardial infarction, coronary artery bypass graft surgery, open heart surgery, or percutaneous transluminal coronary angioplasty within less than 3 months prior to inclusion
* Documentation of >30 premature ventricular complexes per hour, salvos or ventricular tachycardias prior to atrial fibrillation ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal atrial fibrillation scheduled to undergo pulmonary vein isolation
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Ventricular arrhythmias | one year
  Number of patients with premature ventricular complexes, ventricular tachycardias or ventricular fibrillation.

SECONDARY OUTCOMES:
Arrhythmia recurrence | one year
  Number of patients with premature ventricular complexes, ventricular tachycardias or ventricular fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, Prof. Dr., Principal Investigator — Department of Cardiology - Electrophysiology, University Heart Centre
Locations (1):
- Department of Cardiology - Electrophysiology, University Heart Centre, University Hospital Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: PubMed — https://www.ncbi.nlm.nih.gov/pubmed/?term=meyer+jungen+2017
- See also: full version — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5290156/